CLINICAL TRIAL: NCT03520764
Title: A Randomised, Controlled, Double-blind Study to Investigate the Effects of a New Infant Formula on Growth, Safety, and Tolerance in Healthy Term Chinese Infants
Brief Title: To Investigate Effects of a New Infant Formula in Healthy Term Chinese Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Nutricia (Industry)
Collaborators: Nutricia Early Life Nutrition (Shanghai) Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EBB16SI08406
Record Dates: First submitted 2018-03-11; First posted 2018-05-11 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Healthy Infants
MeSH Terms: interventions — Synbiotics; Prebiotics

STUDY DESIGN:
Intervention Model Description: Intervention group: New infant formula with synbiotics; Control group: Standard infant formula with prebiotics
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- New infant formula with synbiotics (Experimental): pHP infant formula with synbiotics (test product)
  Interventions: Dietary Supplement: New infant formula with synbiotics
- Standard infant formula with prebiotics (Active Comparator): Standard (commercial) infant formula with prebiotics (control product)
  Interventions: Dietary Supplement: Standard infant formula with prebiotics
- human milk (No Intervention): Full breastfeeding for at least 17 weeks

INTERVENTIONS:
Dietary Supplement: New infant formula with synbiotics — Infants are fed with synbiotics formula for 17 weeks from the date of enrollment.
  Arms: New infant formula with synbiotics
Dietary Supplement: Standard infant formula with prebiotics — Infants are fed with prebiotics formula for 17 weeks from the date of enrollment.
  Arms: Standard infant formula with prebiotics

SUMMARY:
This study investigates the effects of a new infant formula on growth, safety, and tolerance in healthy term Chinese infants.

Screening starts after the informed consent is obtained. Infants who are less than or equal to 44 days of age and meeting all eligibility criteria will be enrolled into the study. The total duration of the study is around 12 months which includes 8 study visits.

Infants, whose mother has the intention to fully breastfeed her infant at least until 17 weeks of age will be enrolled into the breastfeeding reference group. Infants, whose mother has the intention to fully formula feed her infant as of 44 days of age at the latest, will be randomized to receive either the investigational product or control product until infants reach the age of 17 weeks. After the age of 17 weeks, infants can switch to any feeding and continue be followed up until 12 months of age.

Safety, growth and tolerance parameters will be followed and collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese term infants ≤ 44 days
2. Birth weight within normal range
3. Head circumference within normal range
4. Fully formula fed by the time of randomization OR fully breastfed and with intention to fully breastfeed until 17 weeks of age

Exclusion Criteria:

- The mothers of infants:

1. who are currently participating or will participate in any other (clinical) study involving investigational or marketed products during pregnancy and/or lactation;
2. known to have a significant medical condition that might interfere with the study or known to affect intra-uterine growth, as per investigator's clinical judgement;

   - Parents/Legally acceptable representatives/Caregivers of infants:
3. who are incapable to comply with study protocol

   - Infants:
4. who have to be fed with a special diet other than standard cow's milk based infant formula;
5. known to have current or previous illnesses/conditions which could interfere with the study products or its outcome parameters
6. known or suspected to have an allergic condition towards cow's milk, soy or fish;
7. with any history of, or current participation in any other study involving investigational or marketed products.

Max Age: 44 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 284 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
Weight gain per day from baseline (g/day) | at the age of 17 weeks

SECONDARY OUTCOMES:
Weight gain per day from baseline (g/day) in infant receiving test product compared to breastfed infant. | at the age of 17 weeks
Increment per day from baseline on length (mm/day) | at the age of 17 weeks
Increment per day from baseline on head circumference (mm/day) | at the age of 17 weeks
Increment per day from baseline on mid-upper arm circumference (mm/day) | at the age of 17 weeks
Z-scores of anthropometric parameters from baseline on weight | from baseline until the age of 17 weeks
Z-scores of anthropometric parameters from baseline on length | from baseline until the age of 17 weeks
Z-scores of anthropometric parameters from baseline on head circumference | from baseline until the age of 17 weeks
Z-scores of anthropometric parameters from baseline on mid-upper arm circumference | from baseline until the age of 17 weeks
Effect on incidence, frequency and severity of (serious) adverse events | from baseline until the age of 17 weeks
Parent-reported occurrence of diarrhea | from baseline until the age of 17 weeks
Parent-reported severity of diarrhea | from baseline until the age of 17 weeks
Parent-reported occurrence of constipation | from baseline until the age of 17 weeks
Parent-reported severity of constipation | from baseline until the age of 17 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Peking University 3rd Hospital, Beijing, Beijing Municipality
  - Guangzhou women and Children's Medical Center, Guangzhou, Guangdong
  - Guangdong Province Maternal and Children Hospital, Guangzhou, Guangdong
  - Wuxi Poeple's Hospital, Wuxi, Jiangsu
  - Shanghai Public Health Clinical Research Center, Shanghai, Shanghai Municipality
  - Xin Hua Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Wopereis H, Kakourou A, Liu M, Wu J, Li Z, Zhang L, Tan M, Low JSY, Liu M, Roeselers G, Knol J, Cai W. Restoration of gut microbiota with a specific synbiotic-containing infant formula in healthy Chinese infants born by cesarean section. Eur J Clin Nutr. 2025 Jun;79(6):567-575. doi: 10.1038/s41430-025-01571-8. Epub 2025 Feb 6. PMID 39915586